CLINICAL TRIAL: NCT04171245
Title: Can a Laughter Prescription Improve Psychological Health, Wellbeing, and Sleep in Zayed University Students?
Brief Title: Prescribing Laughter for Sleep and Wellbeing in UAE University Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zayed University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ZU19_064_F
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-10

CONDITIONS: Sleep; Mental Health Wellness
Keywords: Sleep, laughter, well-being, mental health
MeSH Terms: conditions — Laughter; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): One minute laughter prescription 3x a day Tracking sleep using equipment
  Interventions: Other: Laughie laughter prescription; Device: Sleep tracking equipment
- Control (Active Comparator): Tracking sleep using equipment
  Interventions: Device: Sleep tracking equipment

INTERVENTIONS:
Other: Laughie laughter prescription — Creation of a Laughie; laughing with their Laughie 3x a day
  Arms: Experimental
Device: Sleep tracking equipment — Tracking sleep using equipment

SUMMARY:
This study is in line with the UAEs national drive to promote happiness and wellbeing. University students risk impaired psychological health, wellbeing, and sleep due to academic pressures. This research is the first to assess the feasibility of using a laughter prescription to improve psychological health and sleep in Zayed University students. Forty students will be recruited, and randomized to a control or laughter group.

DETAILED DESCRIPTION:
The Laughie is a self created app or tool. It is a one minute recording of the user's joyful laughter on their smartphone. Once recorded, the user uses it by playing back the recording and laughing with it for the duration of the one minute. The Laughie acts as a prompt to guide the one minute of laughter.

In this research the experimental group each record their own Laughie, demonstrated and supported by the PI(s). They are then prescribed to laugh with their Laughie: 3x a day the first week (morning, lunch, and afternoon) and at least 2x a day during the second week. Immediately after using their Laughie they fill in a Laughie checklist to record whether they laughed for the full minute, whether they enjoyed their Laughie, and how they felt afterwards.

This study tracks sleep using wrist actigraphy in the control group (no Laughie prescription) and in the Laughie group. All participants complete one week baseline using sleep watches, and sleep diaries, prior to the Laughie intervention. They all then continue to track their sleep during the intervention. All participants complete WHO Five well-being, PSKI, and HADS pre and post intervention. During the intervention the Laughie participants complete Laughie checklists. All participants are invited for a final interview (the control group about the sleep equipment experience). A follow-up survey is sent to the Laughie group 2 months after their prescription.

ELIGIBILITY:
Inclusion Criteria: Registered Zayed University students, owner of a smartphone -

Exclusion Criteria: Chronic health conditions (cardiovascular disease, respiratory disease, cancer, diabetes), deafness, non-English speakers

-

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-09-26 (Actual); Primary Completion 2020-03-15 (Estimated); Study Completion 2020-04-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility of two-week laughter prescription | 6 months
  Using the Laughie. Evaluate with Laughie checklists and interviews

SECONDARY OUTCOMES:
Assess if subjective sleep outcomes improve | 6 months
  Using PSKI and interviews
Assess if objective sleep outcomes improve | 6 months
  Using wrist actigraphy
Assess if overall well-being improves | 6 months
  Using WHO Five, Laughie checklists, and interviews
Assess if specific aspects of wellbeing improve | 6 months
  Using WHO Five, Laughie checklists, interviews
Assess if mental health improves | 6 months
  Using HADS, interviews

CONTACTS AND LOCATIONS:
Locations (1):
- Zayed University, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonot-Schoupinsky FN, Garip G, Sheffield D, Omar OM, Arora T. Prescribing laughter to ameliorate mental health, sleep, and wellbeing in university students: A protocol for a feasibility study of a randomised controlled trial. Contemp Clin Trials Commun. 2020 Nov 26;20:100676. doi: 10.1016/j.conctc.2020.100676. eCollection 2020 Dec. PMID 33305066